CLINICAL TRIAL: NCT04994483
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, 52-week Study Evaluating the Safety and Efficacy of Simufilam 100 mg Tablets in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Simufilam 100 mg for Mild-to-Moderate Alzheimer's Disease
Acronym: RETHINK-ALZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-125-07
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Intervention Model Description: Approximately 750 patients will be enrolled into the study. All patients will be randomized (1:1) to receive either placebo or 100 mg tablets of simufilam, twice daily, for 52 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized treatments will be assigned by subject numbers in a randomly generated numeric sequence. Randomization (1:1) will be stratified by low or high Mini-Mental State Exam (MMSE; 16-20 and 21-27).
  The randomization code will not be revealed to study subjects, Investigators, clinical staff, study monitors, or the Sponsor until all subjects have completed therapy and the database has been finalized and locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo, supplied by Cassava as coated tablets, and taken twice daily (b.i.d.) for 52 weeks
  Interventions: Drug: Placebo
- Simufilam 100 mg (Experimental): Simufilam 100 mg, supplied by Cassava as coated tablets, and taken b.i.d. for 52 weeks
  Interventions: Drug: Simufilam

INTERVENTIONS:
Drug: Simufilam — Simufilam is a novel drug candidate designed to treat and slow the progression of AD. Simufilam binds with femtomolar affinity to an altered conformation of filamin A that is present in the brain of patients with AD and critical to the toxicity of Aβ42. In this study, simufilam will be given b.i.d. for 52 weeks at a dose of 100 mg.
  Other Names: PTI-125
  Arms: Simufilam 100 mg
Drug: Placebo — Matching placebo given b.i.d. for 52 weeks.
  Arms: Placebo

SUMMARY:
A 52-week safety and efficacy study of simufilam (PTI-125) given twice daily to participants with mild-to-moderate Alzheimer's disease (AD) for 52 weeks. Approximately 750 participants will be randomized (1:1) to receive either placebo or 100 mg tablets of simufilam, twice daily, for 52 weeks. Clinic visits will occur 4 weeks after the baseline visit, and then every 12 weeks until the end of the study. The safety of simufilam, and its efficacy in enhancing cognition and slowing cognitive and functional decline will be evaluated.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety and efficacy of simufilam (PTI-125) in enhancing cognition and slowing cognitive and functional decline following 52-week, repeat-dose oral administration in participants with mild-to-moderate AD. Secondary objectives include the assessment of simufilam's effect on neuropsychiatric symptoms and caregiver burden. A third objective is to investigate the effect of simufilam treatment on plasma biomarkers. A limited number of research sites will be invited to participate in the pharmacokinetic (PK) and plasma biomarker sub-study. Collection of PK samples will enable an exposure-response analysis. Approximately 100 subjects will participate (50 per group). Plasma samples will be collected during the Screening Visit and again at Weeks 28 and 52. Change from Baseline for plasma biomarkers represent additional secondary endpoints.

Safety will be evaluated by adverse event monitoring, vital signs, clinical labs, and the Columbia Suicide Severity Rating Scale at every visit. Subjects will undergo magnetic resonance imaging (MRI) during screening to ensure entry criteria are met (unless recent MRI confirms entry criteria). Resting electrocardiograms will be conducted at Baseline (Study Day 1) and Weeks 4, 28, and 52. A complete physical and neurological examination will be performed at screening, and brief examinations will be performed at all other visits. Weight will be measured during the Screening Period, at Baseline (Study Day 1), and at all other visits.

An independent Data Safety Monitoring Board (DSMB) will meet periodically to review subject safety assessments and determine if dosing may continue. A charter will be developed with specific guidance for the DSMB.

ELIGIBILITY:
Key Inclusion Criteria:

1. Meets National Institute on Aging and Alzheimer's Association Research Framework criteria for individuals in clinical Stage 4 or 5 of the Alzheimer's continuum.
2. Evidence for AD pathophysiology, confirmed either prior to or during screening.
3. MMSE score ≥ 16 and ≤ 27 at screening.
4. Clinical Dementia Rating - Global Score must be 0.5, 1 or 2.
5. If receiving background AD medications, the dosing regimen must be stable for at least 12 weeks prior to randomization. Chronic medications for conditions other than AD (such as depression) must be prescribed at a stable dose for at least 4 weeks prior to screening.
6. The subject has not been a cigarette smoker or chewed tobacco for at least 3 years.
7. Availability of a study partner.
8. Individuals who have participated in a clinical study with an investigational drug targeting the underlying AD process may be permitted to participate in this study.
9. Completed a COVID-19 vaccine primary series ("fully vaccinated") at least 2 weeks prior to randomization or had an unambiguous COVID-19 infection diagnosed more than 3 months before the start of the Screening Period.

Key Exclusion Criteria:

1. A neurologic condition other than AD that significantly contributes to the subject's dementia.
2. Any current primary psychiatric diagnosis other than AD if it is likely to confound cognitive assessment or ability to comply with study procedures.
3. Geriatric Depression Scale (15-item) score > 8. (Note - a subject with a score > 8 may continue in screening if, in the judgment of the Investigator, the elevated score is not attributed to a major depressive episode).
4. Suicidal ideation during the past 3 months or suicidal behavior during the past 12 months.
5. Alcohol or substance use disorder within 2 years of screening.
6. MRI presence of cerebral vascular or other significant pathology.
7. History of transient ischemic attack or stroke within 12 months of screening
8. Seizure within 12 months of screening.
9. Severe head trauma or head trauma considered likely to be contributing to the subject's cognitive impairment.
10. Sleep apnea that is considered likely to be contributing to the subject's cognitive impairment.
11. Insufficiently controlled diabetes mellitus or hypertension.
12. Body mass index < 18.5 or > 37.5.
13. History or diagnosis of clinically significant cardiac disease
14. Currently or previously prescribed/administered aducanumab, lecanemab, or any anti-amyloid monoclonal antibody, more than 2 doses.

Ages: 50 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kupiec, MD, Study Chair — Cassava Sciences
Locations (88):
- United States (74):
  - MDFirst Research, Chandler, Arizona
  - CCT Research - Gilbert Neurology Partners, Gilbert, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - Advanced Research Center, Inc, Anaheim, California
  - Axiom Research, LLC, Colton, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Senior Clinical Trials, Laguna Hills, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Syrentis Clinical Research, Santa Ana, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Colorado Neurological Research Center, PC, Denver, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Topaz Clinical Research, Apopka, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Boynton Beach Medical Research Institute (GMI), Boynton Beach, Florida
  - K2 Medical Research - Clermont, Clermont, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Galiz Research, Hialeah, Florida
  - Infinity Clinical Research - Sunrise, Hollywood, Florida
  - CNS Healthcare - Jacksonville, Jacksonville, Florida
  - Charter Research, Lady Lake, Florida
  - Segal Trials - West Broward Outpatient Site, Lauderhill, Florida
  - ClinCloud, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Central Miami Medical Institute (GMI), Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Luminous Clinical Research, Miami, Florida
  - Quantam Clinical Trials, Miami Beach, Florida
  - South Florida Research Phase I-IV INC, Miami Springs, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of Brandon, LLC (Tampa), Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Premier Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Ascension Via Christi Research, Wichita, Kansas
  - Neuro Medical Clinic of Central Louisiana, LLC, Alexandria, Louisiana
  - Boston Neuro Research Center, North Dartmouth, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - CCT Research - Papillion Research Center, Papillion, Nebraska
  - Advanced Clinical Institute, Inc, West Long Branch, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - Parker Jewish Institute for Health Care & Rehabilitation, New Hyde Park, New York
  - Mid Hudson Medical Research, New Windsor, New York
  - NY Neurology Associates, New York, New York
  - University of Rochester Medical Center - Alzheimer's Disease Care, Research and Education Program, Rochester, New York
  - Five Town Neuroscience Research, Woodmere, New York
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Alzheimer's Memory Center, Matthew, North Carolina
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - NeuroScience Research Center, LLC, Canton, Ohio
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Summit Research Network, LLC, Portland, Oregon
  - Brian Abaluck, LLC, Malvern, Pennsylvania
  - Global Medical Institutes/Scranton Medical Institute - Moosic Division, Moosic, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Palmetto Clinical Research, Summerville, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Senior Adults Specialty Research, Inc, Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Mt. Olympus Medical Research, LLC, Katy, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Green Mountain Research Institute, Inc., Rutland, Vermont
  - Re:Cognition Health, Fairfax, Virginia
  - Memory and Brain Wellness Center at Harborview, Seattle, Washington
- Australia (9):
  - KaRa MINDS, Macquarie Park, New South Wales
  - The University of Queensland, Herston, Queensland
  - Impact Health Pty Ltd., Southport, Queensland
  - Eastern Health, Box Hill, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Canada (5):
  - LMC Clinical Research - London, London, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Q & T Research, Sherbrooke, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Alpha Recherche Clinique, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kupiec JW, Porsteinsson AP, Turner RS, Hendrix S, Mallinckrodt C, Khan A, Cohen I, Liss J, Clarnette R, Park KH, Hernandez AM, Burns LH. Phase 3 randomized clinical trials of simufilam in mild-to-moderate Alzheimer's disease. J Prev Alzheimers Dis. 2026 Jan 1:100469. doi: 10.1016/j.tjpad.2025.100469. Online ahead of print. PMID 41500915

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simufilam 100 mg | Placebo
Started | 403 | 401
Completed | 310 | 325
Not Completed | 93 | 76
Not completed — Adverse Event | 26 | 17
Not completed — Lost to Follow-up | 6 | 10
Not completed — Noncompliance with study drug | 8 | 5
Not completed — Physician Decision | 5 | 0
Not completed — Withdrawal by Subject | 41 | 38
Not completed — Sponsor requests subject to be withdrawn | 2 | 1
Not completed — Met stopping criteria | 1 | 0
Not completed — Randomized in error, not treated | 4 | 3
Not completed — Lack of a reliable study partner | 0 | 1
Not completed — Met MRI exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simufilam 100 mg | Placebo | Total
Number analyzed (Participants) | 403 | 401 | 804
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.72 (7.911) | 74.31 (7.555) | 74.02 (7.737)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 62 | 47 | 109
  65 to 74 years | 126 | 133 | 259
  ≥75 years | 215 | 221 | 436
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 222 | 447
  Male | 178 | 179 | 357
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 51 | 113
  Not Hispanic or Latino | 334 | 341 | 675
  Unknown or Not Reported | 7 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 2 | 10
  Black or African American | 20 | 18 | 38
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  White | 366 | 376 | 742
  Other | 4 | 1 | 5
  Multiple | 1 | 0 | 1
  Not reported | 0 | 1 | 1
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 31 | 21 | 52
  United States | 336 | 355 | 691
  Australia | 36 | 25 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 12-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog12)
Description: The change from baseline to Week 52 in the ADAS-Cog12, a psychometrician-administered battery comprised of several cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Scores range from 0 (best) to 80 (worst).
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 306 | 320
score on a scale | 2.79 (0.363) | 3.19 (0.359)
Statistical Analysis 1: Comparison: Simufilam 100 mg vs Placebo; Test type: Superiority; p = 0.4308, Mixed Models Analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.37 to 0.59]

2. Primary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL)
Description: The change from baseline to Week 52 in the ADCS-ADL, a 23-item study partner questionnaire that covers both basic activities of daily living (ADL) and more complex ADL or instrumental ADL. Scores range from 0 to 78, with a lower score indicating greater severity of functional loss.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 306 | 320
score on a scale | -3.26 (0.442) | -3.76 (0.438)
Statistical Analysis 1: Comparison: Simufilam 100 mg vs Placebo; Test type: Superiority; p = 0.4034, Mixed Models Analysis; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.68 to 1.70]

3. Secondary Outcome: Change From Baseline in the Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: The change from baseline to Week 52 in the iADRS, where scores range from 0 to 146 with lower scores indicating worse performance.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 302 | 317
score on a scale | -5.53 (0.605) | -6.49 (0.598)

4. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory (NPI)
Description: The change from baseline to Week 52 in the NPI, a 12-item study partner interview, which records the frequency and severity of common neuropsychiatric symptoms in dementia, as well as the level of study partner distress due to each of the neuropsychiatric problems. Scores range from 0 to 144, with higher scores indicating more frequent and severe symptoms, and greater levels of partner distress.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 301 | 316
score on a scale | 0.54 (0.588) | 0.90 (0.579)

5. Secondary Outcome: Change From Baseline in the Mini-Mental State Exam (MMSE)
Description: The change from baseline to Week 52 in the MMSE, a set of standardized questions covering several target areas: orientation, registration, attention and calculation, short-term verbal recall, naming, repetition, 3-step command, reading, writing, and visuospatial cognitive assessment. Scores range from 0 to 30, lower scores indicate more severe impairment.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 309 | 324
score on a scale | -1.95 (0.223) | -2.14 (0.221)

6. Secondary Outcome: Change From Baseline in the Clinical Dementia Rating Sum of Boxes (CDR-SB)
Description: The change from baseline to Week 52 in the CDR-SB, which characterizes 6 domains of cognitive and functional performance applicable to AD and related dementias: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Scores for each domain have a minimum of 0 and a maximum of 3, and the 6 domain scores are summed to give the CDR-SB, which has a minimum score of 0 and a maximum score of 18. Higher scores indicate more severe impairment.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 334 | 339
score on a scale | 1.04 (0.138) | 0.85 (0.136)

7. Secondary Outcome: Change From Baseline in the Zarit Burden Interview (ZBI)
Description: The change from baseline to Week 52 in the ZBI, a 22-item study partner questionnaire designed to assess the stress or burden experienced by caregivers of people with dementia. Scores range from 0 to 88, with a higher score indicating greater stress or burden.
Time Frame: Baseline (Study Day 1) to Week 52
Population: Data are from subjects in the Intent-to-treat population (all randomized subjects) who completed the assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 308 | 321
score on a scale | 2.52 (0.556) | 2.30 (0.551)

8. Other Pre Specified Outcome: Changes From Baseline in Plasma Biomarkers
Description: Change from baseline in the following plasma biomarkers of AD pathology, neurodegeneration, and neuroinflammation: phospho-tau217 (P-tau217), glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL), and total tau.
Time Frame: Baseline (Study Day 1) to Week 52
Population: The overall number of participants analyzed is the number of participants who consented to take part in the biomarker analysis substudy and for whom there were baseline values for each biomarker. Plasma samples were not obtained from the whole substudy population at Week 52.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 57 | 62
pg/mL
  P-tau217: number analyzed (Participants) | 45 | 45
  P-tau217 | 1.0 (6.56) | -0.4 (9.77)
  GFAP: number analyzed (Participants) | 45 | 46
  GFAP | 2.0 (57.39) | 40.2 (255.14)
  NfL: number analyzed (Participants) | 45 | 46
  NfL | 69.3 (373.43) | 17.5 (96.73)
  Total tau: number analyzed (Participants) | 45 | 46
  Total tau | 5.5 (35.62) | -2.2 (41.98)

9. Other Pre Specified Outcome: Changes From Baseline in the Plasma SavaDx Biomarker
Description: Change from baseline in SavaDx, a novel plasma biomarker
Time Frame: Baseline (Study Day 1) to Week 52
Population: Change from baseline in SavaDx, a novel plasma biomarker, was included in the protocol as part of the secondary analysis as a biomarker which may have been measured. The final SAP, which postdated the protocol, included the analysis of biomarkers as an exploratory/tertiary endpoint. However, analysis of SavaDx was not conducted due to a sponsor decision and therefore, no results are available.
Arm/Group | Simufilam 100 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 54 weeks after subjects took their first dose of study drug, or until resolution or stabilization of any AEs ongoing at the end of the study.
Description: Data are from the safety population, which included all subjects who received at least 1 dose of study drug.
Arm/Group | Simufilam 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/399 | 3/398
Serious Adverse Events (participants affected / at risk) | 52/399 | 36/398
Other Adverse Events (participants affected / at risk) | 161/399 | 140/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simufilam 100 mg (N=399) | Placebo (N=398)
Hip fracture (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Magnetic resonance imaging hepatobiliary abnormal (Investigations) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simufilam 100 mg (N=399) | Placebo (N=398)
COVID-19 (Infections and infestations) | 29 (29) | 35 (36)
Urinary tract infection (Infections and infestations) | 29 (34) | 27 (35)
Upper respiratory tract infection (Infections and infestations) | 11 (13) | 8 (8)
Headache (Nervous system disorders) | 18 (19) | 11 (14)
Dizziness (Nervous system disorders) | 21 (23) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 30 (38) | 28 (35)
Diarrhoea (Gastrointestinal disorders) | 16 (17) | 16 (16)
Constipation (Gastrointestinal disorders) | 11 (12) | 8 (8)
Nausea (Gastrointestinal disorders) | 10 (11) | 5 (5)
Weight decreased (Investigations) | 6 (6) | 10 (10)
Anxiety (Psychiatric disorders) | 14 (14) | 9 (11)
Depression (Psychiatric disorders) | 10 (10) | 11 (11)
Agitation (Psychiatric disorders) | 9 (9) | 5 (5)
Fatigue (General disorders) | 11 (11) | 11 (11)
Hypertension (Vascular disorders) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and PI must request review and comment of any proposed publication by the sponsor at least 90 days prior to submission of the publication. The sponsor will advise of any information which is confidential information or which may impair the sponsor's ability to obtain patent protection, and has the right to require confidential information or factual errors to be removed, or to delay the proposed publication by an additional 90 days to allow the sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT04994483/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04994483/SAP_001.pdf